CLINICAL TRIAL: NCT04628052
Title: The Effect of Music on Colonoscopy (MUSICOL): A Randomized Controlled Trial
Brief Title: The Effect of Music on Colonoscopy (MUSICOL)
Acronym: MUSICOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively Closed
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Asim Shuja, Assistant Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020-0548
Record Dates: First submitted 2020-06-19; First posted 2020-11-13 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Procedural Anxiety; Colon Polyp
MeSH Terms: conditions — Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental)
  Interventions: Procedure: Colonoscopy
- No-Music (No Intervention)

INTERVENTIONS:
Procedure: Colonoscopy — Music vs. No-Music
  Arms: Music

SUMMARY:
Colonoscopy is an essential tool for diagnostic evaluation for a wide range of gastrointestinal complaints and is considered the gold standard for colorectal cancer screening. This procedure is often associated with patient anxiety both prior to and during the procedure, as well as discomfort,which is managed with procedural sedation.Anticipation of an uncomfortable experience can deter patients from undergoing the procedure despite it being medically indicated. Music has a number of beneficial effects including improving senses of relaxation and well being. Use of music during colonoscopy is inconsistent and there are no society guidelines or recommendations regarding its use. The investigators hypothesize that music will improve the overall patient experience and enhance endoscopist performance.The investigators propose a randomized controlled trial to study effects of music on both the patient experience and endoscopist performance during colonoscopy. Eligible patients will be randomized to two groups: a "music group" and a "no music"control group.Patients in the music group will be asked for their preference of music to be played during their colonoscopy. For patients in the music group, this music will be played in the procedure room during the procedure, while those in the control group will have no music playing. Patient anxiety and pain will be assessed both before and after the procedure.Overall patient experience after the procedure will be assessed on a likert scale. The performance of the endoscopist will be assessed by measuring adenoma detection rate and adenomas per colonoscopy. Additional outcomes to be assessed include total procedure time and amount of sedation required.

DETAILED DESCRIPTION:
Background/Scientific Rationale:

Colorectal cancer is the third most common diagnosed cancer in the United States and is second only to lung cancer in number of deaths. Widespread adoption of colorectal cancer screening has resulted in earlier detection as well as reduction in mortality. Colonoscopy, compared to other methods of screening has additional benefit in its ability to prevent the development of colon cancer through removal of precancerous polyps.Besides it being considered the gold standard for colorectal cancer screening, colonoscopy is an essential tool for diagnostic evaluation for a wide range of gastrointestinal complaints.Despite the proven success of colorectal cancer screening programs and public understanding of its importance, there remains a gap in adherence. In a recent study, about 64% of eligible patients received CRC screening within the past 10 years, which is far behind the "80% by 2018"target. Besides colonoscopy, alternative tools have been developed in an effort to improve adherence to screening including fecal immunochemical testing and fecal DNA testing. However, these tests still have low sensitivity for advanced adenomas of 24% and 42%, respectively, and lack the added benefit of colonoscopy for prevention of development of colon cancer.Patients often experience feelings of anxiety and anticipated discomfort both prior to and during the procedure; one study reported greater than 50% of patients have moderate to severe anxiety about undergoing the procedure. These concerns regarding an anticipated unpleasant experience deter some patients for whom the procedure is indicated from undergoing this valuable test.Sedation is administered during the procedure to alleviate patient discomfort, but this is associated with potential adverse effects, especially if increasing doses are required in response to increased discomfort or anxiety.Sources of patient anxiety about colonoscopy include the necessary bowel preparation,fear of embarrassment, pain, potential complications, sedation, and the potential of a diagnosis of cancer.This anxiety can increase pain perception in patients: a key predictor of pain during colonoscopy is a patient's pre-procedural anxiety level.This anxiety and pain can manifest in the need for increased sedation, increased length of procedure, and reduced patient satisfaction.One way to improve the patient experience that has been investigated is reduced volume bowel preparations. But, prior studies have also suggested that music during a colonoscopy can significantly improve patient satisfaction, reduce anxiety and pain, and reduce the total sedation medication requirement

The performance of gastroenterologists is measured by quality factors such as adenoma detection rate and adenomas per colonoscopy. A number of techniques have been studied to improve these parameters, including use of colonoscope caps and second looks on the right side of the colon and right-sided retroflexion. Additionally, prior studies have suggested improvement from music being played in the endoscopy suite. An intervention that is inexpensive and without adverse effects that can potentially improve the patient experience and as a consequence hypothetically adherence to screening programs, and improve endoscopist performance, would be expected to be widely adopted. Yet, use of music during colonoscopy is inconsistent and there are no society guidelines or recommendations regarding its use. Potential reasons for this include a sense of a lack of adequate body of evidence and inconsistency in the method of administration.The investigators aim to provide more convincing data to support or refute the benefit of music during colonoscopy to aid the decision on whether routinely offering music during the procedure should be considered a standard of care.

Objectives/Aims:

The investigators' aim is to assess whether playing music during a colonoscopy procedure improves the patient experience and willingness to undergo the procedure again(measured on a Likert scale), improves endoscopist performance (as measured by adenoma detection rate and time to reach cecum), and reduces the mean dose of sedatives required during the procedure (both midazolam and fentanyl).Secondary endpoints include reduction in pain,total procedure time, and withdrawal time.The delay between the time the procedure was scheduled for and the time the procedure actually commenced will also be measured, as long delays are a not uncommon occurrence that can separately negatively impact the patient experience and therefore this variable maybe used for post-hoc analysis. The investigators anticipate the study to take place over the course of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Outpatient
* Undergoing colonoscopy for screening, surveillance, or diagnostic purposes
* Procedure is to be performed solely by an attending gastroenterologist
* Sedation plan is moderate sedation (midazolam, fentanyl, and/or diphenhydramine administered by RN)

Exclusion Criteria:

* Age < 18 and > 80
* Inpatients
* Deafness or hearing loss requiring use of hearing aids
* Patient is prescribed and taking opiate pain medications or benzodiazepine anxiety medications
* Previous history of colon cancer
* Previous history of colon resection
* History of incomplete or aborted colonoscopy procedures
* Participation of an anesthesia professional for administration of monitored anesthesia care of general anesthesia
* ASA PS Classification > 4
* Double procedures (EGD & Colonoscopy)
* A gastroenterology fellow will be participating in the procedure
* Endoscopist cancels the colonoscopy before scope insertion (most commonly due to believing the prep is inadequate or a contraindication identified)
* Minors, and non-English speaking subjects will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Anxiety Score | Up to 1 hour
  Will be using PROMIS anxiety short forms. Patients will be asked if in the past 7 days, they felt anxious or fearful or worried or unable to focus or nervous or uneasy or tense. They will have to choose one option like Never or Rarely or Sometimes or Often or Always.
Dose of Sedative required | Up to 3 hours
Level of Pain | Change from baseline pain level at 2 hours
  Pain will be measured using a 'Likert Scale' on a scale from 0 to 10, 0 being no pain and 10 being the worse possible pain.
Willingness to undergo procedure in future | Upto 3 hours
  Patient willingness to undergo procedure in future will be measure using a '5-point Likert scale' on a scale from 1 to 5, 1 means 'I would never do this procedure again' while 5 means 'I would do it again without any hesitation'.

SECONDARY OUTCOMES:
Total procedure time | Upto 2 hours
  Total time for completion of the procedure, starting from insertion of the scope till the scope is out from the colon.
Time to reach cecum | Upto 1 hour
  Time taken from insertion of the colonoscope in rectum till it reaches the cecum
Withdrawal time | Upto 1 hour
  Time taken from the start of inspection of cecum till the withdrawal of the scope from rectum
Adenoma detection rate | Upto 2 hours
  Number of screening colonoscopies in which one or more adenomas are detected, divided by the total number of screening colonoscopies.
Adenomas per colonoscopy | Upto 2 hours
  Number of detected adenomas divided by the total number of screening colonoscopies.

CONTACTS AND LOCATIONS:
Overall Officials: Asim Shuja, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Berkowitz Z, Zhang X, Richards TB, Nadel M, Peipins LA, Holt J. Multilevel Small-Area Estimation of Colorectal Cancer Screening in the United States. Cancer Epidemiol Biomarkers Prev. 2018 Mar;27(3):245-253. doi: 10.1158/1055-9965.EPI-17-0488. PMID 29500250
- [Background] Song LL, Li YM. Current noninvasive tests for colorectal cancer screening: An overview of colorectal cancer screening tests. World J Gastrointest Oncol. 2016 Nov 15;8(11):793-800. doi: 10.4251/wjgo.v8.i11.793. PMID 27895817
- [Background] Yang C, Sriranjan V, Abou-Setta AM, Poluha W, Walker JR, Singh H. Anxiety Associated with Colonoscopy and Flexible Sigmoidoscopy: A Systematic Review. Am J Gastroenterol. 2018 Dec;113(12):1810-1818. doi: 10.1038/s41395-018-0398-8. Epub 2018 Nov 1. PMID 30385831
- [Background] Hsueh FC, Chen CM, Sun CA, Chou YC, Hsiao SM, Yang T. A Study on the Effects of a Health Education Intervention on Anxiety and Pain During Colonoscopy Procedures. J Nurs Res. 2016 Jun;24(2):181-9. doi: 10.1097/jnr.0000000000000112. PMID 26551213
- [Background] Bashiri M, Akcali D, Coskun D, Cindoruk M, Dikmen A, Cifdaloz BU. Evaluation of pain and patient satisfaction by music therapy in patients with endoscopy/colonoscopy. Turk J Gastroenterol. 2018 Sep;29(5):574-579. doi: 10.5152/tjg.2018.18200. PMID 30260780